CLINICAL TRIAL: NCT00643201
Title: A Safety and Efficacy Trial Evaluating the Use of Apixaban in the Treatment of Symptomatic Deep Vein Thrombosis and Pulmonary Embolism
Brief Title: Efficacy and Safety Study of Apixaban for the Treatment of Deep Vein Thrombosis or Pulmonary Embolism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV185-056; EUDRACT: 2007-007867-25
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Enoxaparin; Warfarin; apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Active Comparator): apixaban: tablets, oral, 10 milligram (mg) tablets, twice daily, for 7 days followed by apixaban 5 mg, twice daily, 6 months.
  Interventions: Drug: Enoxaparin; Drug: warfarin; Drug: Placebo for apixaban
- Enoxaparin + Warfarin (Experimental): Enoxaparin: solution, subcutaneous, 1 mg/kg Q12h until international normalized ratio (INR) ≥2.
  Interventions: Drug: Placebo for enoxaparin; Drug: Placebo for warfarin; Drug: apixaban

INTERVENTIONS:
Drug: Enoxaparin — solution, subcutaneous, 1 mg/kg Q12h until International normalized ratio (INR) ≥2.
  Arms: Apixaban
Drug: warfarin — tablets, oral, dosing to target INR range between 2.0 - 3.0, once daily, 6 months
  Other Names: Coumadin; BMS-565793
  Arms: Apixaban
Drug: Placebo for apixaban — tablets, oral, 10 mg tablets, twice daily, for 7 days followed by placebo for apixaban 5 mg tablets, twice daily, 6 months
  Arms: Apixaban
Drug: Placebo for enoxaparin — solution, subcutaneous, 1 mg/kg Q12h until sham INR ≥2.
  Arms: Enoxaparin + Warfarin
Drug: Placebo for warfarin — tablets, oral, dosing to target sham INR range between 2.0 - 3.0, once daily, 6 months
  Arms: Enoxaparin + Warfarin
Drug: apixaban — tablets, oral, 10 mg tablets, twice daily, for 7 days followed by apixaban 5 mg, twice daily, 6 months
  Other Names: BMS-562247
  Arms: Enoxaparin + Warfarin

SUMMARY:
The purpose of this study is to evaluate the effects of an investigational blood thinner, apixaban, in preventing venous thromboembolic (VTE) recurrence or death in patients with deep vein thrombosis (DVT) or pulmonary embolism (PE)

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Clinical diagnosis of DVT or PE

Exclusion Criteria:

* Contraindications for enoxaparin or warfarin
* Active bleeding or high risk for serious bleeding
* Short life expectancy
* Uncontrolled high blood pressure
* Significantly impaired kidney or liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5614 (Actual)
Dates: Start 2008-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (307):
- United States (73):
  - Alabama Clinical Therapeutics, Llc, Birmingham, Alabama
  - Horizon Research Group, Inc., Mobile, Alabama
  - Fort Smith Lung Center, Fort Smith, Arkansas
  - University Of Arkansas For Medical Sciences, Little Rock, Arkansas
  - Beaver Medical Group, Banning, California
  - University Of California San Francisco-Fresno, Fresno, California
  - University Of California, Davis Medical Center, Sacramento, California
  - Chest Medicine & Critical Care Medical Gr. Inc., San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Harbor Ucla Medical Center, Torrance, California
  - New West Physicians, Golden, Colorado
  - Drogue Medical, Llc, Wheat Ridge, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Dept Of Internal Med, Sect Of Pulmonary & Critical Care Med, New Haven, Connecticut
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Bay Pines Va Healthcare Systems, Bay Pines, Florida
  - Daniel G. Lorch, Jr, Md, Cpi, Brandon, Florida
  - Research Alliance, Inc., Clearwater, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Pasadena Center For Medical Research, St. Petersburg, Florida
  - Tampa Clinical Research, Tampa, Florida
  - Office Of Michele S. Maholtz Md, Vero Beach, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Atlanta Pulmonary Group, Atlanta, Georgia
  - Atlanta Institute For Medical Research, Inc, Decatur, Georgia
  - Chatham Hospitalists, Savannah, Georgia
  - Gateway Cardiology. P.C, Jerseyville, Illinois
  - West Suburban Medical Center, Oak Park, Illinois
  - Infectious Disease Of Indiana Psc, Carmel, Indiana
  - Heartland Vascular Medicine And Surgery, Windsor Heights, Iowa
  - Kentucky Lung Clinic, Hazard, Kentucky
  - Univ. Of Kentucky Dept. Of Surgery, Lexington, Kentucky
  - Research Integrity, Llc, Owensboro, Kentucky
  - Pen Bay Medical Center, Rockport, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Medstar Research Health Institute, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mississippi Medical Research, Llc, Picayune, Mississippi
  - University Of Missouri-Columbia, Columbia, Missouri
  - Veterans Affairs Medical Center, Kansas City, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - St. John'S Mercy Medical Center, St Louis, Missouri
  - Mercury Street Medical Group, Pllc, Butte, Montana
  - Great Falls Clinic, Llp, Great Falls, Montana
  - Internal Medical Associates Of Grand Island, P.C, Grand Island, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Pulmonary & Critical Care Services, Pc, Albany, New York
  - Kaleida Health System, Buffalo, New York
  - Richmond University Medical Center, Staten Island, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Wilmington Medical Research, Wilmington, North Carolina
  - Clinical Trials Of America, Inc., Winston-Salem, North Carolina
  - Altru Health System Clinic, Grand Forks, North Dakota
  - Huron Hospital, Cleveland, Ohio
  - Remington Davis Inc., Columbus, Ohio
  - Oregon Health Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Kore Cv Research, Jackson, Tennessee
  - Primecare Medical Group, Houston, Texas
  - Cancer Care Centers Of South Texas, San Antonio, Texas
  - University Of Utah Medical Center, Salt Lake City, Utah
  - Lake Washington Vascular, Pllc, Bellevue, Washington
  - Franciscan Research Center, Tacoma, Washington
- Argentina (5):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution, Corrientes, Corrientes Province
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
- Australia (14):
  - Local Institution, Garran, Australian Capital Territory
  - Local Institution, Concord, New South Wales
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Lismore, New South Wales
  - Local Institution, Randwick, New South Wales
  - Local Institution, Herston, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Hobart, Tasmania
  - Local Institution, Box Hill, Victoria
  - Local Institution, Clayton, Victoria
  - Local Institution, Ringwood East, Victoria
  - Local Institution, Windsor, Victoria
  - Local Institution, Perth, Western Australia
- Austria (3):
  - Local Institution, Graz
  - Local Institution, Innsbruck
  - Local Institution, Vienna
- Brazil (11):
  - Local Institution, Belo Horizonte - Mg, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Rio Janeiro, Rio de Janeiro
  - Local Institution, Port Alegre, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Botucatu, São Paulo
  - Local Institution, Liberdade, São Paulo
  - Local Institution, São Bernardo do Campo, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (13):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Saint John, New Brunswick
  - Local Institution, Hamilton, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Waterloo, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Saint-Jérôme, Quebec
- Chile (4):
  - Local Institution, Punta Arenas, Magallanes Antartica
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Independencia, Santiago Metropolitan
  - Local Institution, Santiago, Santiago Metropolitan
- China (7):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Wuhan, Hubei
  - Local Institution, Shengyang, Liaoning
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Xi'an
- Czechia (9):
  - Local Institution, Hradec Králové
  - Local Institution, Kladno
  - Local Institution, Litomyšl
  - Local Institution, Městec Králové
  - Local Institution, Ostrava
  - Local Institution, Ostrava Vitkovice
  - Local Institution, Prague
  - Local Institution, Ústí nad Labem
  - Local Institution, Ústí nad Orlicí
- Denmark (7):
  - Local Institution, Arhus C
  - Local Institution, Hellerup
  - Local Institution, Herning
  - Local Institution, Hilleroed
  - Local Institution, Horsens
  - Local Institution, Næstved
  - Local Institution, Silkeborg
- France (17):
  - Local Institution, Angers
  - Local Institution, Arras
  - Local Institution, Besançon
  - Local Institution, Clamart
  - Local Institution, Clermont-Ferrand
  - Local Institution, Dijon
  - Local Institution, Grenoble
  - Local Institution, Langres
  - Local Institution, Le Kremlin-Bicêtre
  - Local Institution, Lille
  - Local Institution, Limoges
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pierre-Bénite
  - Local Institution, Saint-Priest-en-Jarez
  - Local Institution, Toulouse
  - Local Institution, Vernon
- Germany (12):
  - Local Institution, Berlin
  - Local Institution, Bochum
  - Local Institution, Cologne
  - Local Institution, Dortmund
  - Local Institution, Dresden
  - Local Institution, Frankfurt
  - Local Institution, Göttingen
  - Local Institution, Karlsbad
  - Local Institution, Ludwigshafen
  - Local Institution, Mannheim
  - Local Institution, Munich
  - Local Institution, München
- Hong Kong (2):
  - Local Institution, Pokfulman
  - Local Institution, Shatin, N.T
- Hungary (7):
  - Local Institution, Budapest
  - Local Institution, Gyula
  - Local Institution, Kecskemét
  - Local Institution, Miskolc
  - Local Institution, Mosonmagyaróvár
  - Local Institution, Székesfehérvár
  - Local Institution, Zalaegerszeg
- India (12):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Gurgaon, Haryana
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Bengaluru, Karnataka
  - Local Institution, Manipal, Karnataka
  - Local Institution, Pune, Maharashtra
  - Local Institution, Mohali, Punjab
  - Local Institution, Ludhiana, Tagore Nagar
  - Local Institution, Chennai, Tamil Nadu
  - Local Institution, Bangalore
  - Local Institution, Pune
- Israel (14):
  - Local Institution, Tiberias, Lower Galillee
  - Local Institution, Afula
  - Local Institution, Ashkelon
  - Local Institution, Hadera
  - Local Institution, Haifa
  - Local Institution, Holon
  - Local Institution, Jerusalem
  - Local Institution, Kfar Saba
  - Local Institution, Nahariya
  - Local Institution, Petah Tikva
  - Local Institution, Rehovot
  - Local Institution, Safed
  - Local Institution, Tel Aviv
  - Local Institution, Tel Litwinsky
- Italy (16):
  - Local Institution, Bologna
  - Local Institution, Castelfranco Veneto (Tv)
  - Local Institution, Chieti Scalo
  - Local Institution, Cosenza
  - Local Institution, Milan
  - Local Institution, Padua
  - Local Institution, Palermo
  - Local Institution, Pavia
  - Local Institution, Piacenza
  - Local Institution, Pisa
  - Local Institution, Reggio Emilia
  - Local Institution, Rome
  - Local Institution, Rozzano (Mi)
  - Local Institution, San Daniele Del Friuli (Ud)
  - Local Institution, Vicenza
  - Local Institution, Vittorio Veneto (Tv)
- Malaysia (4):
  - Local Institution, Kuala Lumpur, Kuala Lumpur
  - Local Institution, Malacca, Melaka
  - Local Institution, Ipoh, Perak
  - Local Institution, George Town, Pulau Pinang
- Mexico (8):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Durango, Durango
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, León, Guanajuato
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Xalapa, Veracruz
- Norway (8):
  - Local Institution, Ålesund
  - Local Institution, Fredrikstad
  - Local Institution, Gjettum
  - Local Institution, Gjøvik
  - Local Institution, Hamar
  - Local Institution, Oslo
  - Local Institution, Trondheim
  - Local Institution, Tynset
- Poland (11):
  - Local Institution, Bialystok
  - Local Institution, Bydgoszcz
  - Local Institution, Gdansk
  - Local Institution, Gdynia
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Poznan
  - Local Institution, Przeworsk
  - Local Institution, Szczecin
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Portugal (3):
  - Local Institution, Coimbra
  - Local Institution, Guarda
  - Local Institution, Lisbon
- Local Institution, San Juan, Puerto Rico
- Romania (3):
  - Local Institution, Baia Mare
  - Local Institution, Bucharest
  - Local Institution, Târgu Mureş
- Russia (10):
  - Local Institution, Arkhangelsk
  - Local Institution, Chelyabinsk
  - Local Institution, Kazan'
  - Local Institution, Moscow
  - Local Institution, Novosibirsk
  - Local Institution, Rostov-on-Don
  - Local Institution, Ryazan
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Yaroslavl
- Local Institution, Singapore, Singapore
- South Africa (10):
  - Local Institution, Bioemfontein, Free State
  - Local Institution, Centurion, Gauteng
  - Local Institution, Parktown, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Pietermaritzburg, KwaZulu-Natal
  - Local Institution, Bellville, Western Cape
  - Local Institution, George, Western Cape
  - Local Institution, Somerset West, Western Cape
  - Local Institution, Worcester, Western Cape
- South Korea (2):
  - Local Institution, Busan
  - Local Institution, Seoul
- Spain (8):
  - Local Institution, Torrevieja, Alicante
  - Local Institution, Getafe
  - Local Institution, L'Hospitalet de Llobregat
  - Local Institution, León
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Mourente
  - Local Institution, Tarragona
- Ukraine (11):
  - Local Institution, Chernihiv
  - Local Institution, Dnipropetrovsk
  - Local Institution, Donetsk
  - Local Institution, Ivano-Frankivsk
  - Local Institution, Kharkiv
  - Local Institution, Kyiv
  - Local Institution, Lviv
  - Local Institution, Odesa
  - Local Institution, Ternopil
  - Local Institution, Vinnytsia
  - Local Institution, Zaporizhzhia
- Local Institution, Livingston, West Lothian, United Kingdom

REFERENCES:
- [Derived] Jamieson MJ, Byon W, Dettloff RW, Crawford M, Gargalovic PS, Merali SJ, Onorato J, Quintero AJ, Russ C. Apixaban Use in Obese Patients: A Review of the Pharmacokinetic, Interventional, and Observational Study Data. Am J Cardiovasc Drugs. 2022 Nov;22(6):615-631. doi: 10.1007/s40256-022-00524-x. Epub 2022 May 16. PMID 35570249
- [Derived] Cohen AT, Pan S, Byon W, Ilyas BS, Taylor T, Lee TC. Efficacy, Safety, and Exposure of Apixaban in Patients with High Body Weight or Obesity and Venous Thromboembolism: Insights from AMPLIFY. Adv Ther. 2021 Jun;38(6):3003-3018. doi: 10.1007/s12325-021-01716-8. Epub 2021 Apr 22. PMID 33890242
- [Derived] Cohen AT, Agnelli G, Buller HR, Gallus A, Raskob GE, Sanders P, Thompson J, Weitz JI. Characteristics and Outcomes in Patients with Venous Thromboembolism Taking Concomitant Anti-Platelet Agents and Anticoagulants in the AMPLIFY Trial. Thromb Haemost. 2019 Mar;119(3):461-466. doi: 10.1055/s-0038-1676983. Epub 2019 Jan 16. PMID 30650446
- [Derived] Liu X, Johnson M, Mardekian J, Phatak H, Thompson J, Cohen AT. Apixaban Reduces Hospitalizations in Patients With Venous Thromboembolism: An Analysis of the Apixaban for the Initial Management of Pulmonary Embolism and Deep-Vein Thrombosis as First-Line Therapy (AMPLIFY) Trial. J Am Heart Assoc. 2015 Dec 1;4(12):e002340. doi: 10.1161/JAHA.115.002340. PMID 26627879
- [Derived] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Masiukiewicz U, Pak R, Thompson J, Raskob GE, Weitz JI; AMPLIFY Investigators. Oral apixaban for the treatment of acute venous thromboembolism. N Engl J Med. 2013 Aug 29;369(9):799-808. doi: 10.1056/NEJMoa1302507. Epub 2013 Jul 1. PMID 23808982
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant, first visit: 27 August 2008; Last participant, last visit: 12 March 2013.
Pre-assignment Details: 5614 enrolled, 5395 randomized; Reasons for non-randomization: 173 did not meet inclusion/exclusion criteria; 12 withdrew consent; 5 had clinical reason to continue current treatment; 3 administrative reason by sponsor; 1 death; 1 adverse event (AE); 24 other reasons. 1 site (5 patients) excluded from analysis due to unconfirmed accuracy of data.
Groups:
- Apixaban: apixaban: tablets, oral, 10 milligram (mg) tablets, twice daily, for 7 days followed by apixaban 5 mg, twice daily, 6 months.
  Placebo for enoxaparin: solution, subcutaneous, 1milligram per kilogram (mg/kg) every 12 hours until sham international normalized ratio (INR) greater than, equal to ( ≥) 2.
  Placebo for warfarin: tablets, oral, dosing to target sham INR range between 2.0 - 3.0, once daily, 6 months
- Enoxaparin + Warfarin: Enoxaparin: solution, subcutaneous, 1 mg/kg Q12h until INR ≥2.
  Warfarin: tablets, oral, dosing to target INR range between 2.0 - 3.0, once daily, 6 months
  Placebo for apixaban: tablets, oral, 10 mg tablets, twice daily, for 7 days followed by placebo for apixaban 5 mg tablets, twice daily, 6 months
Period: Randomized, Completed 6 Months of Study
Arm/Group | Apixaban | Enoxaparin + Warfarin
Started | 2691 (15 participants were randomized to treatment but not treated.) | 2704 (15 participants were randomized to treatment but not treated.)
Completed | 2314 | 2291
Not Completed | 377 | 413
Not completed — Death | 20 | 26
Not completed — Adverse Event | 150 | 182
Not completed — Withdrawal by Subject | 49 | 49
Not completed — Lost to Follow-up | 14 | 14
Not completed — Poor or non-compliance | 20 | 23
Not completed — Pregnancy | 3 | 2
Not completed — Fails to meet inclusion/exclusion | 13 | 9
Not completed — Administrative reason | 1 | 1
Not completed — Other | 107 | 107
Period: Completed Study Follow Up
Arm/Group | Apixaban | Enoxaparin + Warfarin
Started | 2617 | 2639
Completed | 2547 (Of 70 who did not complete follow up: 7 completed treatment; 63 discontinued treatment) | 2560 (Of 79 who did not complete follow up: 3 completed treatment, 76 discontinued treatment)
Not Completed | 70 | 79
Not completed — Death | 28 | 34
Not completed — Withdrawal by Subject | 23 | 29
Not completed — Lost to Follow-up | 18 | 16
Not completed — non-specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Enoxaparin + Warfarin | Total
Number analyzed (Participants) | 2691 | 2704 | 5395
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (15.98) | 56.7 (16.01) | 56.9 (16.00)
Age, Customized [Number; unit: participants]
  Less than (<) 65 | 1729 | 1762 | 3491
  65 to < 75 | 560 | 570 | 1130
  Greater than, equal to (>=) 75 | 402 | 372 | 774
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1122 | 1106 | 2228
  Male | 1569 | 1598 | 3167
Race/Ethnicity, Customized [Number; unit: participants] — Ethnicity was not collected outside of the United States.
  participants
    White | 2218 | 2243 | 4461
    Black or African American | 106 | 98 | 204
    American Indian or Alaska Native | 6 | 2 | 8
    Asian | 227 | 226 | 453
    Other Race | 89 | 85 | 174
    Race Not Reported | 45 | 50 | 95
    Hispanic or Latino | 20 | 18 | 38
    Not Hispanic or Latino | 367 | 380 | 747
    Ethnicity Not Reported | 2304 | 2306 | 4610
Region of Enrollment [Number; unit: participants]
  Portugal | 10 | 9 | 19
  United States | 387 | 398 | 785
  Hong Kong | 2 | 1 | 3
  Spain | 56 | 51 | 107
  Ukraine | 213 | 211 | 424
  Israel | 162 | 163 | 325
  Russian Federation | 178 | 174 | 352
  Italy | 167 | 169 | 336
  India | 101 | 99 | 200
  France | 140 | 149 | 289
  Malaysia | 0 | 2 | 2
  Australia | 56 | 64 | 120
  Denmark | 69 | 72 | 141
  South Africa | 70 | 77 | 147
  China | 113 | 114 | 227
  Korea, Republic of | 2 | 2 | 4
  Austria | 40 | 39 | 79
  Czech Republic | 140 | 134 | 274
  Hungary | 145 | 128 | 273
  Mexico | 59 | 57 | 116
  Canada | 147 | 152 | 299
  Argentina | 17 | 16 | 33
  Poland | 60 | 59 | 119
  Brazil | 77 | 81 | 158
  Singapore | 5 | 5 | 10
  Romania | 33 | 41 | 74
  Norway | 40 | 32 | 72
  Germany | 202 | 205 | 407
Qualifying index Venous Thromboembolic Embolism [Number; unit: participants] — Both the 2004 and 2008 American College of Chest Physicians (ACCP) recommendations for treatment of venous thromboembolic events (VTE) were used during this study and recommendations were consistent. Participants with provoked and unprovoked index events were summarized. For unprovoked events in participants with certain risk factors and medical conditions, such as cancer, an idiopathic event, presence of pro-thrombotic genotype, or presence of a marker indicative of an increased risk of recurrent thromboembolism treatment for 6 months or longer is supported by the ACCP guidelines.
  participants
    Provoked Index VTE | 272 | 272 | 544
    Unprovoked Index VTE | 2416 | 2429 | 4845
    Not Reported | 3 | 3 | 6
Index Event Classification [Number; unit: participants] — Participants with events of either deep vein thrombosis (DVT) or pulmonary embolism (PE) were enrolled. If a participant had both DVT and PE, the participant was classified to PE. Each participant was counted once in a category but could be counted in more than one category. An Independent Central Adjudication Committee (ICAC) reviewed participants in a blinded manner. The ICAC included a chairman and independent reviewers who were physicians with experience in vascular medicine and thrombosis. The ICAC adjudicated all index events (proximal DVT and/or PE).
  participants
    Proximal DVT | 1778 | 1814 | 3592
    PE | 913 | 890 | 1803
    Adjudicated Proximal DVT | 1749 | 1783 | 3532
    Adjudicated PE | 930 | 906 | 1836

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adjudicated Composite of Symptomatic, Recurrent Venous Thromboembolism (VTE) or VTE-Related Death During 6 Months of Treatment
Description: VTE: nonfatal deep vein thrombosis (DVT) or nonfatal pulmonary embolism (PE). All events were adjudicated by an ICAC blinded to treatment. DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate (proportion of participants): n/N (n=number of participants with observation; N=total number of efficacy evaluable participants). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early). Composite endpoint: events at any time from randomization until end of intended treatment, regardless whether drug treatment was received. All randomized participants with a non-missing primary endpoint were summarized. Missing endpoint = outcomes which could not be documented on or after study Day 154. Participants were categorized to the assigned group regardless of the treatment actually received (intent-to-treat).
Time Frame: Day 1 to Week 24 + 2 Days or 355 days (Discontinued Early)
Population: All randomized participants with a non-missing primary endpoint (n/N: 59/2609; 71/2635, in apixaban, enoxaparin/warfarin, respectively). Intent-to-treat population. Confidence interval (CI) for event rate calculated based on the Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Apixaban: Apixaban: tablets, oral, 10 mg tablets, twice daily, for 7 days followed by apixaban 5 mg, twice daily, 6 months
  Placebo for enoxaparin: solution, subcutaneous, 1 mg/kg Q12h until sham INR ≥2.
  Placebo for warfarin: tablets, oral, dosing to target sham INR range between 2.0 - 3.0, once daily, 6 months
- Enoxaparin + Warfarin: Enoxaparin: solution, subcutaneous, 1 mg/kg Q12h until INR ≥2
  warfarin: tablets, oral, dosing to target INR range between 2.0 - 3.0, once daily, 6 months
  Placebo for apixaban: tablets, oral, 10 mg tablets, twice daily, for 7 days followed by placebo for apixaban 5 mg tablets, twice daily, 6 months
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2609 | 2635
proportion of participants | 0.0226 [0.0169 to 0.0283] | 0.0269 [0.0208 to 0.0331]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Hypothesis that apixaban was non-inferior to enoxaparin/warfarin therapy in preventing the recurrence of VTE (nonfatal DVT or nonfatal PE)/VTE-related death; Test type: Non-Inferiority or Equivalence — Statistical Testing: non-inferiority tested at 1-sided α=0.025 with margin of 1.8. Demonstration of non-inferiority using both relative risk (RR) (margin = 1.8) and risk difference (RD) (margin = 0.035) were required to achieve the primary objective; p < 0.0001, Yanagawa-Tango-Hiejima — This is the first test in a sequential testing sequence. p-value calculated based on the Yanagawa-Tango-Hiejima test stratified by index event strata for non-inferiority. Tested at 1-sided α=0.025; For a successful trial; rejection of the null hypotheses for both RR and RD was required; Risk Ratio (RR) = 0.8390, 95% CI 2-sided [0.5965 to 1.1802]
Statistical Analysis 2: Comparison: Apixaban vs Enoxaparin + Warfarin; Hypothesis that apixaban was non-inferior to enoxaparin/warfarin therapy in preventing the recurrence of VTE (nonfatal DVT or nonfatalPE)/VTE-related death as measured by risk difference; Test type: Non-Inferiority or Equivalence — Statistical Testing; non-inferiority tested at 1-sided α=0.025. If non-inferiority demonstrated for both RR and RD, the primary objective was achieved; p < 0.0001, Yanagawa-Tango-Hiejima — Yanagawa-Tango-Hiejima test statistic for risk difference (RD); Risk Difference (RD) = -0.0044, 95% CI 2-sided [-0.0128 to 0.0040]
Statistical Analysis 3: Comparison: Apixaban vs Enoxaparin + Warfarin; Hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint. Inferential testing required demonstration of non-inferiority using both RR and RD plus demonstration of superiority for major bleeding; Test type: Superiority or Other; p = 0.3128, Cochran-Mantel-Haenszel — Tested at 2-sided α=0.05 significance. Further inferential statistical testing halted due to failure to reject the null hypothesis of equivalence for VTE/VTE-related death; Relative risk, CI, and p-value were calculated based on CMH test stratified by index event strata; Risk Ratio (RR) = 0.8390, 95% CI 2-sided [0.5965 to 1.1802]

2. Secondary Outcome: Incidence of Adjudicated Composite of Recurrent Symptomatic Venous Thromboembolism (VTE) or All-Cause Death
Description: VTE included: nonfatal DVT or nonfatal PE. All events were adjudicated by an ICAC blinded to treatment. DVT was assessed by compression ultrasound and/or venography; PE was assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate (proportion of participants with event) calculated as n/N (n=number of participants with observation; N=total number of efficacy evaluable participants). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early). Composite endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received, ie intent to treat (ITT) principle. Each participant scored as having an event only if they experienced one or more of the elements of the composite. Participants with missing endpoint information excluded.
Time Frame: Day 1 up to 24 Weeks + 2 Days or 355 Days (Discontinued Early)
Population: All randomized participants with non-missing secondary endpoint (n/N: 84/2609; 104/2635, in apixaban, enoxaparin/warfarin arms, respectively). Participants categorized to assigned arm, regardless of treatment actually received. Intent to Treat principle. Confidence interval (CI) for event rate calculated based on Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Apixaban: Apixaban: tablets, oral, 10 mg tablets, twice daily, for 7 days followed by apixaban 5 mg, twice daily, 6 months
  Placebo for enoxaparin: solution, subcutaneous, 1 mg/kg Q12h until sham INR ≥2
  Placebo for warfarin: tablets, oral, dosing to target sham INR range between 2.0 - 3.0, once daily, 6 months
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2609 | 2635
proportion of participants | 0.0322 [0.0254 to 0.0390] | 0.0395 [0.0320 to 0.0469]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; p = 0.1554, Cochran-Mantel-Haenszel — The test was stratified by index event strata using alpha=0.05 level of significance. Analysis was performed on the secondary efficacy dataset; there was no imputation of missing data; Nominal p-value is reported; Risk Ratio (RR) = 0.8151, 95% CI 2-sided [0.6146 to 1.0812]

3. Secondary Outcome: Incidence of Adjudicated Composite of Recurrent Symptomatic VTE or Cardiovascular (CV)-Related Death
Description: VTE included: nonfatal DVT or nonfatal PE. All events were adjudicated by an ICAC blinded to treatment. DVT was assessed by compression ultrasound and/or venography; PE was assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate (proportion of participants with event) calculated as n/N (n=number of participants with observation; N=total number of efficacy evaluable participants, participants with missing endpoint information excluded). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early). Composite endpoint included events at any time from randomization until end of the intended treatment period, regardless whether drug treatment was received, ie, ITT principle. Each participant scored as having an event only if the participant experienced one or more of the elements of the composite.
Time Frame: Day 1 up to 24 Weeks + 2 Days or 355 Days (Discontinued Early)
Population: All randomized participants with non-missing secondary endpoint (n/N: 61/2609; 77/2635, in apixaban, enoxaparin/warfarin arms, respectively). Participants categorized to assigned arm, regardless of treatment actually received. Intent to Treat principle. CI for event rate calculated based on Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2609 | 2635
proportion of participants | 0.0234 [0.0176 to 0.0292] | 0.0292 [0.0228 to 0.0357]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; p = 0.1848, Cochran-Mantel-Haenszel — The test was stratified by index event strata using alpha=0.05 level of significance. . Nominal p-value is reported; Analysis was performed on the secondary efficacy dataset; there was no imputation of missing data; Risk Ratio (RR) = 0.7994, 95% CI 2-sided [0.5737 to 1.1137]

4. Secondary Outcome: Incidence of Adjudicated Composite of Recurrent Symptomatic VTE or VTE-related Death or Major Bleeding
Description: VTE included: nonfatal DVT or nonfatal PE. All events were adjudicated by an ICAC blinded to treatment. DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Major bleeding defined by International Society on Thrombosis and Haemostasis: acute, clinically overt bleeding associated with decrease in hemoglobin (Hgb) of 2 g/dL or more or bleeding leading to transfusion or bleeding in a critical site or bleeding that is fatal . Event rate (proportion of participants with event): n/N (n=number of participants with observation; N=Total number of participants, excluding those with missing endpoint and including those not in the efficacy evaluable population with a bleeding event that occurred during treatment period. Events included regardless of whether or not participant received treatment, ie, ITT principle
Time Frame: Day 1 up to 24 Weeks + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants in each randomized arm, excluded those with missing endpoint and included those not in the efficacy evaluable population with bleeding event which occurred during treatment (n/N: 73/2610; 118/2635). Confidence interval (CI) for event rate calculated based on Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2610 | 2635
proportion of participants | 0.0280 [0.0216 to 0.0343] | 0.0448 [0.0369 to 0.0527]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel — The test was stratified by index event strata using alpha=0.05 level of significance. Nominal p-value is reported; Risk Ratio (RR) = 0.6236, 95% CI 2-sided [0.4682 to 0.8306]

5. Secondary Outcome: Incidence of Adjudicated Composite of Recurrent Symptomatic VTE, Myocardial Infarction, Stroke, CV-related Death, Clinically Relevant Non-major (CRNM) Bleeding or Major Bleeding
Description: VTE=Nonfatal DVT or nonfatal PE adjudicated by ICAC blinded to treatment. DVT: compression ultrasound and/or venography; PE: spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Major Bleeding = acute, clinically overt bleeding: decrease in Hgb of 2 g/dL or more or bleeding leading to transfusion or bleeding in a critical site or fatal bleeding. CRNM = acute clinically overt bleeding: compromising hemodynamics, leading to hospitalization, hematoma, epistasis >5 minutes or repetitive, gingival bleeding, hematuria, macroscopic gastrointestinal hemorrhage, rectal blood loss, hemoptysis. n/N (n=number of participants with observation; N=Total number of participants, excluding those with missing endpoint and including those not in the efficacy evaluable population with a bleeding event that occurred during treatment period). Events included regardless of whether or not treatment was received (ITT).
Time Frame: Day 1 up to 24 Weeks + 2 Days or 355 Days (Discontinued Early)
Population: Total number participants in each treatment group, excluded those with missing endpoint and included those not in the efficacy evaluable population with bleeding event which occurred during treatment (n/N: 183/2617; 333/2641). Events included as per ITT principle. CI for event rate calculated based on Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2617 | 2641
proportion of participants | 0.0699 [0.0602 to 0.0797] | 0.1261 [0.1134 to 0.1387]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The test was stratified by index event strata using alpha=0.05 level of significance. Nominal p-value is reported; Risk Ratio (RR) = 0.5532, 95% CI 2-sided [0.4658 to 0.6569]

6. Secondary Outcome: Incidence of Adjudicated Symptomatic Nonfatal Deep Vein Thrombosis (DVT) During the Intended Treatment Period
Description: DVT adjudicated by an ICAC blinded to treatment. DVT evaluated by: compression ultrasound and/or venography. Includes events that occurred during the intended treatment period, regardless of whether the participant received study medication, intent to treat principle (ITT). Event rate (proportion of participants with event): n/N (n=number of participants with observation; N=Total number of participants, excluding those with missing endpoint). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early).
Time Frame: Day 1 up to 24 Weeks + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants in each randomized arm (ITT), excluding those with missing endpoint (n/N: 22/2608; 35/2633). CI for event rate calculated based on Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2608 | 2633
proportion of participants | 0.0084 [0.0049 to 0.0119] | 0.0133 [0.0089 to 0.0177]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.6347, 95% CI 2-sided [0.3735 to 1.0787] — Relative Risk and CI was calculated based on CMH test stratified by index event strata

7. Secondary Outcome: Incidence of Adjudicated Symptomatic Nonfatal Pulmonary Embolism (PE) During the Intended Treatment Period
Description: PE adjudicated by an ICAC blinded to treatment. PE: spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Includes events that occurred during the intended treatment period, regardless of whether the participant received study medication (ITT principle). Event rate (proportion of participants with event): n/N (n=number of participants with observation; N=Total number of participants, excluding those with missing endpoint). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early).
Time Frame: Day 1 to Week 24 + + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants in each randomized arm (ITT), excluding those with missing endpoint (n/N: 27/2606; 25/2632). CI for event rate calculated based on Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2606 | 2632
proportion of participants | 0.0104 [0.0065 to 0.0142] | 0.0095 [0.0058 to 0.0132]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.0935, 95% CI 2-sided [0.6363 to 1.8793] — Relative Risk and CI was calculated based on CMH test stratified by index event strata

8. Secondary Outcome: Incidence of Adjudicated Venous Thromboembolism (VTE)-Related Death During the Intended Treatment Period
Description: VTE-related death included: DVT-related death or PE-related death. All events were adjudicated by an ICAC blinded to treatment. DVT was assessed by compression ultrasound and/or venography; PE was assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate (proportion of participants with event) calculated as n/N (n=number of participants with observation; N=total number of participants in respective treatment groups excluding participants with missing endpoint information). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early). Includes events that occur during the intended treatment period regardless of whether or not the participant received study medication (ITT principle).
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants in respective treatment groups excluding participants with missing endpoint information. (n/N: 12/2608; 16/2630). CI for event rate calculated based on Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2608 | 2630
proportion of participants | 0.0046 [0.0020 to 0.0072] | 0.0061 [0.0031 to 0.0091]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.7521, 95% CI 2-sided [0.3560 to 1.5889] — Relative Risk and CI was calculated based on CMH test stratified by index event strata

9. Secondary Outcome: Incidence of Cardiovascular (CV)-Related Death Including VTE-related Death During the Intended Treatment Period
Description: VTE-related death included: DVT-related death or PE-related death. All events were adjudicated by an ICAC blinded to treatment. DVT assessed by compression ultrasound and/or venography; PE assessed by spiral computed tomography scanning, pulmonary angiography, and/or ventilation/perfusion lung scan. Event rate (proportion of participants with event) calculated as n/N (n=number of participants with observation; N=total number of participants in respective treatment groups excluding participants with missing endpoint information). Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early). Includes events that occur during the intended treatment period regardless of whether or not the participant received study medication (ITT principle).
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants in respective groups excluding those with missing endpoint information (n/N: 15/2608; 23/2630). CI for event rate calculated based on Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2608 | 2630
proportion of participants | 0.0058 [0.0028 to 0.0087] | 0.0087 [0.0052 to 0.0123]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.6539, 95% CI 2-sided [0.3419 to 1.2508] — Relative Risk and CI was calculated based on CMH test stratified by index event strata

10. Secondary Outcome: Incidence of All-Cause Death During the Intended Treatment Period
Description: Intended treatment period: longer of the dosing period plus 2 days (completed treatment) or 355 days (discontinued early). Includes events that occurred during the intended treatment period, regardless of whether the participant received study medication (ITT principle). Event rate (proportion of participants with event): n/N (n=number of participants with observation; N=Total number of participants, excluding those with missing endpoint information).
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants excluding those with missing endpoint (n/N: 41/2608; 52/2630). Events included regardless of whether or not participant received treatment, ie, ITT principle. CI for event rate calculated based on Wald asymptotic confidence limits.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2608 | 2630
proportion of participants | 0.0157 [0.0109 to 0.0205] | 0.0198 [0.0145 to 0.0251]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.7934, 95% CI 2-sided [0.5287 to 1.1906] — Relative Risk and CI was calculated based on CMH test stratified by index event strata

11. Secondary Outcome: Incidence of Adjudicated Major Bleeding During the Treatment Period in Treated Participants
Description: All events were adjudicated by an ICAC blinded to treatment. Bleeding defined by International Society on Thrombosis and Haemostasis: Major Bleeding: acute, clinically overt bleeding: decrease in hemoglobin (hgb) of 2 g/dL or more or bleeding leading to transfusion or bleeding in a critical site or fatal bleeding. Event rate (proportion of participants with event): n/N (n=number of participants with observation; N=Total number of participants in respective treatment group (all participants who received at least one dose of study drug). Participants were categorized to the treatment group to which they were assigned unless incorrect study treatment was received throughout the study, in which case the participant was categorized according to the treatment received.
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants receiving at least one dose of study drug n/N: 15/2676; 49/2689, in apixaban and enoxaparin/warfarin groups, respectively. CI for event rate calculated based on Wald asymptotic confidence limits. Participants were categorized according to the actual treatment received.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2676 | 2689
proportion of participants | 0.0056 [0.0028 to 0.0084] | 0.0182 [0.0132 to 0.0233]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Hypothesis: apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint. As per the hierarchical statistical testing cascade, inferential testing for adjudicated major bleeding occurred because non-inferiority for VTE/VTE-related death (Primary efficacy endpoint) was demonstrated earlier. Rejection of the null hypothesis for equivalence for major bleeding allowed inferential testing for superiority of VTE/VTE-related death; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — p-value calculated on the CMH test stratified by index event strata; Risk Ratio (RR) = 0.3070, 95% CI 2-sided [0.1728 to 0.5452] — Relative risk and CI were calculated based on CMH test stratified by index event strata

12. Secondary Outcome: Incidence of Adjudicated Major/CRNM Bleeding During the Treatment Period in Treated Participants
Description: Major Bleeding = acute, clinically overt bleeding: decrease in hemoglobin of 2 g/dL or more, or bleeding leading to transfusion, or bleeding in a critical site, or fatal bleeding. CRNM = acute clinically overt bleeding: compromising hemodynamics, leading to hospitalization, hematoma, epistasis >5 minutes or repetitive, gingival bleeding, hematuria, macroscopic gastrointestinal hemorrhage, rectal blood loss, hemoptysis. Minor =: All acute clinically overt bleeding events not meeting the criteria for either major bleeding or CRNM. All events were adjudicated by an ICAC blinded to treatment. Total bleeding = any of major, or CRNM, or minor bleeding. Event rate (proportion of participants with event): n/N (n=number of participants with observation; N=Total number of treated (received at least 1 dose of study drug).
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants receiving at least one dose of study drug n/N: 115/2676; 261/2689, in apixaban and enoxaparin/warfarin groups, respectively. CI for event rate calculated based on Wald asymptotic confidence limits. Participants were categorized according to the actual treatment received.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2676 | 2689
proportion of participants | 0.0430 [0.0353 to 0.0507] | 0.0971 [0.0859 to 0.1083]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint. Inferential testing was not conducted because the null hypothesis pertaining to superiority for VTE/VTE-related death was not rejected; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Tested at 2-sided alpha=0.05 significance; Nominal p-value is reported; Risk Ratio (RR) = 0.4410, 95% CI 2-sided [0.3566 to 0.5453] — Relative Risk and CI was calculated based on CMH test stratified by index event strata

13. Secondary Outcome: Incidence of Adjudicated Clinically Relevant Non Major (CRNM) Bleeding During the Treatment Period in Treated Participants
Description: Bleeding defined by International Society on Thrombosis and Haemostasis: CRNM defined as acute clinically overt bleeding: compromising hemodynamics, leading to hospitalization, hematoma, epistasis >5 minutes or repetitive, gingival bleeding, hematuria, macroscopic gastrointestinal hemorrhage, rectal blood loss, hemoptysis. All events were adjudicated by an ICAC blinded to treatment. Event rate (proportion of participants with event): calculated as n/N (n=number of participants with observation; N=Total number of participants in respective treatment group (all participants who received at least one dose of study drug). Participants were categorized to the treatment group to which they were assigned unless incorrect study treatment was received throughout the study, in which case the participant was categorized according to the treatment received.
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants receiving at least one dose of study drug n/N: 103/2676; 215/2689, in apixaban and enoxaparin/warfarin groups, respectively. CI for event rate calculated based on Wald asymptotic confidence limits. Participants were categorized according to the actual treatment received.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2676 | 2689
proportion of participants | 0.0385 [0.0312 to 0.0458] | 0.0800 [0.0697 to 0.0902]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Tested at 2-sided alpha=0.05 significance; Nominal p-value is reported; Risk Ratio (RR) = 0.4793, 95% CI 2-sided [0.3815 to 0.6022] — Relative Risk and CI was calculated based on CMH test stratified by index event strata

14. Secondary Outcome: Incidence of Adjudicated Minor Bleeding During the Treatment Period in Treated Participants
Description: Bleeding defined by International Society on Thrombosis and Haemostasis: Minor bleeding: all acute clinically overt bleeding events not meeting the criteria for either major bleeding or CRNM. All events wre adjudicated by an ICAC blinded to treatment. Event rate (proportion of participants) calculated as n/N (n=number of participants with observation; N=Total number of participants in respective treatment group (all participants who received at least one dose of study drug). Participants were categorized to the treatment group to which they were assigned unless incorrect study treatment was received throughout the study, in which case the participant was categorized according to the treatment received.
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants receiving at least one dose of study drug n/N: 313/2676; 505/2689, in apixaban and enoxaparin/warfarin groups, respectively. CI for event rate calculated based on Wald asymptotic confidence limits. Participants were categorized according to the actual treatment received.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2676 | 2689
proportion of participants | 0.1170 [0.1048 to 0.1291] | 0.1878 [0.1730 to 0.2026]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Tested at 2-sided alpha=0.05 significance; Nominal p-value is reported; Risk Ratio (RR) = 0.6182, 95% CI 2-sided [0.5432 to 0.7034] — Relative Risk and CI was calculated based on CMH test stratified by index event strata

15. Secondary Outcome: Incidence of Adjudicated Total Bleeding During the Treatment Period in Treated Participants
Description: Bleeding defined by International Society on Thrombosis and Haemostasis: Total Bleeding defined as any of major, CRNM, or minor bleeding. All events were adjudicated by an ICAC blinded to treatment. Event rate (proportion of participants with event): n/N (n=number of participants with observation; N=Total number of participants in respective treatment group (all participants who received at least one dose of study drug). Participants were categorized to the treatment group to which they were assigned unless incorrect study treatment was received throughout the study, in which case the participant was categorized according to the treatment received.
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: Total number of participants receiving at least one dose of study drug n/N: 402/2676; 676/2689, in apixaban and enoxaparin/warfarin groups, respectively. CI for event rate calculated based on Wald asymptotic confidence limits. Participants were categorized according to the actual treatment received.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2676 | 2689
proportion of participants | 0.1502 [0.1367 to 0.1638] | 0.2514 [0.2350 to 0.2678]
Statistical Analysis 1: Comparison: Apixaban vs Enoxaparin + Warfarin; Exploratory hypothesis of apixaban therapy being superior to enoxaparin/warfarin therapy for the adjudicated endpoint; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Tested at 2-sided alpha=0.05 significance; Nominal p-value is reported; Risk Ratio (RR) = 0.5937, 95% CI 2-sided [0.5318 to 0.6629] — Relative Risk and CI was calculated based on CMH test stratified by index event strata

16. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Bleeding AEs, Discontinuations Due to AEs and Death During the Treatment Period in Treated Participants
Description: Treated Participants: all who received at least 1 dose of study drug. Participants categorized to the treatment group to which they were assigned unless incorrect study treatment was received throughout the study, in which case the participant was categorized according to treatment received. Included all SAEs and AEs with onset from first dose to last dose + 2 days (for AEs) or + 30 days (for SAEs); note; bleeding AEs and SAEs from first dose to last dose + 2 days included. Discontinuations due to AE included all AEs/SAEs from first dose until drug was discontinued. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: First dose to last dose of 24 Weeks + 2 days (AEs) or + 30 days (SAEs) or until drug discontinued
Population: Total number of participants receiving at least one dose of study drug. Participants were categorized according to the actual treatment received.
Measure: Number; unit: participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2676 | 2689
participants
  AE | 1795 | 1923
  SAE | 417 | 410
  Bleeding AE or SAE | 415 | 695
  Discontinued Due to AE or SAE | 162 | 199
  Death | 37 | 44

17. Secondary Outcome: Number of Treated Participants With Marked Abnormalities in Hematology Laboratory Tests
Description: Lower limit of normal (LLN). Upper limit of normal (ULN). Pre-therapy (PreRx). Absolute (Abs) neutrophil count, bands + neutrophils (ANC). Cells per microliter (c/µL). Grams per deciliter (g/dL). Cells per Liter (c/L). Millimeter (MM). White blood cells: < 0.75*LLN, > 1.25*ULN; Hemoglobin: <= 11.5 g/dL (males), <= 9.5 g/dL (females); Hematocrit: <= 37% (males), <= 32% (females); Erythrocytes: <0.75*10^6 c/µL*PreRx; Platelet count: < 75*10^9 c/L, > 700*10^9 c/L; ANC: < 1.00*10^3 c/µL; Abs eosinophils: > 0.750*10^3 c/µL; Abs Basophils: > 400/MM^3; Abs Monocytes> 2000/MM^3; Abs Lymphocytes: < 0.750*10*3 c/ µL, > 7.5*10^3 c/ µL.
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: N=Treated participants who received at least one dose of study drug and had non-missing laboratory measurements.
Measure: Number; unit: participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2599 | 2593
participants
  Erthrocytes Low (N=2599, 2593) | 23 | 17
  Hematocrit Low (N=2588, 2587) | 26 | 20
  Hemoglobin Low (N=2599, 2593) | 96 | 101
  Platelet Count Low (N=2594, 2589) | 23 | 13
  Leukocytes Low (N=2528, 2519) | 41 | 41
  Leukocytes High (N=2528, 2519) | 26 | 15
  Absolute Basophils High (N=2594,2589) | 1 | 2
  Absolute Eosinophils High (N=2594,2589) | 84 | 79
  Absolute Lyphocytes Low (N=2594,2589) | 94 | 76
  Absolute Lyphocytes High (N=2594,2589) | 4 | 3
  Absolute Monocytes High (N=2594,2589) | 1 | 2
  Absolute Neutrophils Low (N=2594,2589) | 9 | 20

18. Secondary Outcome: Number of Treated Participants With Marked Abnormalities in Electrolyte Laboratory Tests
Description: Bicarbonate milliequivalents/Liter (mEq/L) Low/High: < 0.75*LLN or > 1.25*ULN, or if pre-dose < LLN then use < 0.75*pre-dose or > ULN if pre-dose > ULN then use > 1.25*pre-dose or < LLN; Serum Calcium mg/dL Low/High: < 0.8*LLN or > 1.2*ULN, or if pre-dose < LLN then use < 0.75*pre-dose or > ULN if pre-dose > ULN then use > 1.25*pre-dose or < LLN; Serum Chloride mEq/L: < 0.9*LLN or > 1.1*ULN, or if pre-dose < LLN then use < 0.9*pre-dose or > ULN if pre-dose > ULN then use > 1.1*pre-dose or < LLN; Serum Potassium mEq/L: < 0.9*LLN or > 1.1*ULN, or if pre-dose < LLN then use < 0.9*pre-dose or > ULN if pre-dose > ULN then use > 1.1*pre-dose or < LLN; Serum Sodium mEq/L: < 0.95*LLN or > 1.05*ULN, or if pre-dose < LLN then use < 0.95*pre-dose or > ULN if pre-dose > ULN then use > 1.05*pre-dose or < LLN.
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: N=Treated participants who received at least one dose of study drug and had non-missing laboratory measurements.
Measure: Number; unit: participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2601 | 2596
participants
  Bicarbonate Low (N=2600,2593) | 44 | 31
  Bicarbonate High (N=2600,2593) | 17 | 11
  Total Calcium Low (N=2601,2596) | 3 | 10
  Total Calcium High (N=2601,2596) | 12 | 11
  Chloride Low Total Calcium Low (N=2601,2596) | 5 | 3
  Chloride Low Total Calcium High (N=2601,2596) | 0 | 1
  Potassium Low (N=2601,2596) | 26 | 22
  Potassium High (N=2601,2596) | 19 | 22
  Sodium Low (N=2601,2596) | 10 | 6
  Sodium Low (N=2601,2596) | 4 | 4

19. Secondary Outcome: Number of Treated Participants With Marked Abnormalities in Kidney and Liver Function Laboratory Tests
Description: Blood urea nitrogen (BUN), milligrams/deciliter (mg/dL), units per liter (U/L). BUN mg/dL High: > 1.5*ULN; Creatinine mg/dL: > 1.5*ULN; Alanine aminotransferase (ALT) U/L: > 3*ULN; Aspartate aminotransferase (AST) U/L: > 3*ULN; Alkaline phosphatase U/L: > 2*ULN; Bilirubin Direct mg/dL: > 1.5*ULN; Bilirubin Total mg/dL: > 2*ULN.
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: N=Treated participants who received at least one dose of study drug and had non-missing laboratory measurements.
Measure: Number; unit: participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2601 | 2598
participants
  BUN High (N=517, 523) | 2 | 7
  Creatinine High (N=2601, 2596) | 47 | 37
  ALT High (N=2601, 2598) | 52 | 145
  ALP High (N=2601, 2598) | 35 | 27
  AST High (N=2601, 2598) | 40 | 40
  Direct Bilirubin High (N=2601, 2593) | 28 | 21
  Total Bilirubin High (N=2601, 2597) | 8 | 7

20. Secondary Outcome: Number of Treated Participants With Marked Abnormalities in Creatine Kinase, Uric Acid, and Total Protein Laboratory Tests
Description: Creatine kinase High: >5*ULN Units/Liter (U/L); Total Protein High/Low: < 0.9 *LLN or > 1.1*ULN, or if pre-dose < LLN then use 0.9* pre-dose or > ULN if pre-dose > ULN then use 1.1 *pre-dose or <LLN; Uric acid High: > 1.5* ULN, or if pre-dose > ULN then use > 2 *pre-dose.
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: N=Treated participants who received at least one dose of study drug and had non-missing laboratory measurements.
Measure: Number; unit: participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 2601 | 2596
participants
  Creatine Kinase High (N=2601, 2596) | 20 | 24
  Uric Acid High (N=2601, 2596) | 6 | 3
  Total Protein Low (N=2601, 2596) | 15 | 16
  Total Protein High (N=2601, 2596) | 0 | 0

21. Secondary Outcome: Number of Treated Participants With Marked Abnormalities in Urinalysis Laboratory Tests
Description: All tests in urine: Glucose: If missing pre-dose use ≥ 2, or if value ≥ 4, or if pre-dose = 0 or 0.5 use ≥ 2, or if pre-dose = 1 use ≥ 3, or if pre-dose = 2 or 3 use ≥ 4; Protein: If missing pre-dose use ≥ 2, or if value ≥ 4, or if pre-dose = 0 or 0.5 use ≥ 2, or if pre-dose = 1 use ≥ 3, or if pre-dose = 2 or 3 use ≥ 4; Blood: If missing pre-dose use ≥ 2, or if value ≥ 4, or if pre-dose = 0 or 0.5 use ≥ 2, or if pre-dose = 1 use ≥ 3, or if pre-dose = 2 or 3 use ≥ 4; Leukocyte esterase: If missing pre-dose use ≥ 2, or if value ≥ 4, or if pre-dose = 0 or 0.5 use ≥ 2, or if pre-dose = 1 use ≥ 3, or if pre-dose = 2 or 3 use ≥ 4;Red blood cells (RBC): If missing pre-dose use ≥ 2, or if value ≥ 4, or if pre-dose = 0 or 0.5 use ≥ 2, or if pre-dose = 1 use ≥ 3, or if pre-dose = 2 or 3 use ≥ 4; White blood cells (WBC): If missing pre-dose use ≥ 2, or if value ≥ 4, or if pre-dose = 0 or 0.5 use ≥ 2, or if pre-dose = 1 use ≥ 3, or if pre-dose = 2 or 3 use ≥ 4.
Time Frame: Day 1 to Week 24 + 2 Days or 355 Days (Discontinued Early)
Population: N=Treated participants who received at least one dose of study drug and had non-missing laboratory measurements.
Measure: Number; unit: participants
Arm/Group | Apixaban | Enoxaparin + Warfarin
Number analyzed (Participants) | 1685 | 1719
participants
  Blood in Urine High (N=2289, 2273) | 85 | 127
  Glucose in Urine High (N=2289, 2273) | 46 | 31
  Leukocyte Esterase in Urine High (N=2289, 2273) | 105 | 102
  Protein in Urine High (N=2289, 2273) | 41 | 50
  RBC + WBC in Urine High (N=1685, 1719) | 359 | 361
  RBC in Urine High (N=1293, 1389) | 111 | 140
  WBC in Urine High (N=1354, 1361) | 274 | 263

ADVERSE EVENTS:
Time Frame: Day 1 up to 24 Weeks + 2 Days or 355 Days (for those participants who discontinued early)/
Groups:
- Enoxaparin/Warfarin: Enoxaparin: solution, subcutaneous, 1 mg/kg Q12h until INR ≥2
  warfarin: tablets, oral, dosing to target INR range between 2.0 - 3.0, once daily, 6 months
  Placebo for apixaban: tablets, oral, 10 mg tablets, twice daily, for 7 days followed by placebo for apixaban 5 mg tablets, twice daily, 6 months
Arm/Group | Apixaban | Enoxaparin/Warfarin
Serious Adverse Events (participants affected / at risk) | 417/2676 | 410/2689
Other Adverse Events (participants affected / at risk) | 1014/2676 | 1207/2689
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=2676) | Enoxaparin/Warfarin (N=2689)
ANAEMIA (Blood and lymphatic system disorders) | 6 | 4
ANAEMIA MEGALOBLASTIC (Blood and lymphatic system disorders) | 1 | 0
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 0 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 1
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
HILAR LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 5 | 2
ANGINA PECTORIS (Cardiac disorders) | 3 | 1
ANGINA UNSTABLE (Cardiac disorders) | 1 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 6 | 7
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 | 0
ATRIAL THROMBOSIS (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 1
BRADYCARDIA (Cardiac disorders) | 1 | 1
CARDIAC ARREST (Cardiac disorders) | 2 | 1
CARDIAC FAILURE (Cardiac disorders) | 5 | 8
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 5 | 2
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 0 | 2
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 5
DILATATION VENTRICULAR (Cardiac disorders) | 0 | 1
INTRACARDIAC THROMBUS (Cardiac disorders) | 1 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 3
PALPITATIONS (Cardiac disorders) | 1 | 0
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 1 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0
PRINZMETAL ANGINA (Cardiac disorders) | 1 | 0
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 | 0
VENTRICULAR HYPOKINESIA (Cardiac disorders) | 0 | 1
SICKLE CELL ANAEMIA WITH CRISIS (Congenital, familial and genetic disorders) | 0 | 1
INNER EAR DISORDER (Ear and labyrinth disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 1
RETINAL HAEMORRHAGE (Eye disorders) | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 2
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 1 | 2
ABDOMINAL WALL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 1 | 0
COLONIC POLYP (Gastrointestinal disorders) | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DIAPHRAGMATIC HERNIA (Gastrointestinal disorders) | 0 | 1
DIVERTICULUM (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
DUODENITIS (Gastrointestinal disorders) | 0 | 1
DUODENOGASTRIC REFLUX (Gastrointestinal disorders) | 0 | 1
DYSPEPSIA (Gastrointestinal disorders) | 1 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1
ENTERITIS (Gastrointestinal disorders) | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRIC POLYPS (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 2
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 8 | 14
GASTROINTESTINAL HYPOMOTILITY (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROLITHIASIS (Gastrointestinal disorders) | 1 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 2 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 2
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 1
MELAENA (Gastrointestinal disorders) | 1 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 0 | 1
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0
PANCREATITIS RELAPSING (Gastrointestinal disorders) | 0 | 1
PERITONEAL CYST (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 3
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
TONGUE OEDEMA (Gastrointestinal disorders) | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 | 0
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
ASTHENIA (General disorders) | 1 | 2
AXILLARY PAIN (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 3 | 4
DEATH (General disorders) | 4 | 2
DEVICE OCCLUSION (General disorders) | 1 | 0
HERNIA OBSTRUCTIVE (General disorders) | 1 | 0
MULTI-ORGAN DISORDER (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 3 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 9 | 6
OEDEMA PERIPHERAL (General disorders) | 3 | 3
PELVIC MASS (General disorders) | 0 | 1
PYREXIA (General disorders) | 4 | 1
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 2 | 3
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 2 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 2 | 2
CHOLESTASIS (Hepatobiliary disorders) | 0 | 1
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 | 1
HEPATIC CYST (Hepatobiliary disorders) | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 2
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 1
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 | 0
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 | 1
AUTOIMMUNE DISORDER (Immune system disorders) | 0 | 1
BEHCET'S SYNDROME (Immune system disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 2 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 0
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 | 1
ABSCESS INTESTINAL (Infections and infestations) | 0 | 1
ABSCESS LIMB (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 4 | 2
BRONCHITIS BACTERIAL (Infections and infestations) | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 3
CARDIAC VALVE VEGETATION (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 6 | 3
CELLULITIS ORBITAL (Infections and infestations) | 1 | 0
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0
CYSTITIS (Infections and infestations) | 1 | 0
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 1 | 2
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 3 | 2
GASTROENTERITIS (Infections and infestations) | 2 | 3
GENITAL HERPES (Infections and infestations) | 1 | 0
GROIN ABSCESS (Infections and infestations) | 0 | 1
HELICOBACTER GASTRITIS (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0
INFECTED SKIN ULCER (Infections and infestations) | 1 | 1
INFECTION (Infections and infestations) | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0
LUNG ABSCESS (Infections and infestations) | 1 | 0
LUNG INFECTION (Infections and infestations) | 1 | 0
MASTOIDITIS (Infections and infestations) | 1 | 0
MYCOBACTERIAL INFECTION (Infections and infestations) | 1 | 0
MYELITIS (Infections and infestations) | 1 | 0
OROPHARYNGEAL CANDIDIASIS (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 2 | 1
PERINEAL ABSCESS (Infections and infestations) | 0 | 1
PERITONITIS (Infections and infestations) | 1 | 0
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 16 | 12
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 | 1
PURULENT PERICARDITIS (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 1 | 2
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
SEPSIS (Infections and infestations) | 5 | 5
SEPTIC SHOCK (Infections and infestations) | 3 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
TONSILLITIS (Infections and infestations) | 0 | 1
TUBERCULOSIS (Infections and infestations) | 1 | 0
TULARAEMIA (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 8 | 3
UROSEPSIS (Infections and infestations) | 4 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 1
VULVAL ABSCESS (Infections and infestations) | 0 | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 2 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 2 | 0
DRUG ADMINISTRATION ERROR (Injury, poisoning and procedural complications) | 1 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 1
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
FACE INJURY (Injury, poisoning and procedural complications) | 1 | 0
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
INCORRECT DOSE ADMINISTERED (Injury, poisoning and procedural complications) | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 15 | 11
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
PERIPHERAL ARTERIAL REOCCLUSION (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
RENAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 0 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 2
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 1
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
COAGULATION TIME PROLONGED (Investigations) | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 1
HEPATIC ENZYME INCREASED (Investigations) | 1 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 3 | 7
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 3
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 4 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
FRACTURE MALUNION (Musculoskeletal and connective tissue disorders) | 0 | 1
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
LIGAMENT DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 6 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 2
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 2 | 0
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 0 | 1
PSEUDARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 1
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 | 1
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
BENIGN OVARIAN TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
BLADDER PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BONE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BRAIN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
BREAST CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CERVIX NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
ENDOCRINE NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ESSENTIAL THROMBOCYTHAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GALLBLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GASTRIC CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GASTROINTESTINAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
MALIGNANT PERITONEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO ABDOMINAL CAVITY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC CARCINOMA OF THE BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
METASTATIC RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OESOPHAGEAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ONCOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
PANCREATIC CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PANCREATIC CARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PANCREATIC NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PARAPROTEINAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PELVIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
POLYCYTHAEMIA VERA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RECTOSIGMOID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
TESTIS CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
TUMOUR ULCERATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 2 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 | 2
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 | 1
COMA (Nervous system disorders) | 1 | 0
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 1 | 2
ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
GRAND MAL CONVULSION (Nervous system disorders) | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 2 | 1
HEADACHE (Nervous system disorders) | 0 | 2
ISCHAEMIC STROKE (Nervous system disorders) | 5 | 5
LACUNAR INFARCTION (Nervous system disorders) | 1 | 0
MIGRAINE (Nervous system disorders) | 1 | 0
MULTIPLE SCLEROSIS (Nervous system disorders) | 2 | 0
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 | 1
NEURALGIA (Nervous system disorders) | 1 | 0
NEURITIS (Nervous system disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0
PARAPLEGIA (Nervous system disorders) | 1 | 0
PERONEAL NERVE PALSY (Nervous system disorders) | 1 | 0
POLYNEUROPATHY (Nervous system disorders) | 1 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 1
SCIATICA (Nervous system disorders) | 2 | 3
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 2
SYNCOPE (Nervous system disorders) | 3 | 3
THALAMIC INFARCTION (Nervous system disorders) | 1 | 0
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 | 3
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 | 0
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 5 | 2
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 | 1
ALCOHOL ABUSE (Psychiatric disorders) | 0 | 1
ALCOHOLISM (Psychiatric disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 3 | 2
APATHY (Psychiatric disorders) | 1 | 0
BIPOLAR DISORDER (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 1
DEPRESSION (Psychiatric disorders) | 2 | 3
DEPRESSION SUICIDAL (Psychiatric disorders) | 1 | 0
MENTAL DISORDER (Psychiatric disorders) | 1 | 0
PANIC ATTACK (Psychiatric disorders) | 0 | 2
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 0
TIC (Psychiatric disorders) | 1 | 0
GLOMERULONEPHRITIS CHRONIC (Renal and urinary disorders) | 0 | 1
GLOMERULONEPHRITIS MEMBRANOPROLIFERATIVE (Renal and urinary disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 5 | 13
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 0 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 3 | 1
OLIGURIA (Renal and urinary disorders) | 1 | 0
RENAL COLIC (Renal and urinary disorders) | 0 | 1
RENAL CYST HAEMORRHAGE (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 3 | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 | 3
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0
URINARY BLADDER HAEMORRHAGE (Renal and urinary disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 | 1
ENDOMETRIAL HYPERTROPHY (Reproductive system and breast disorders) | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 2 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 1
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 2 | 2
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
ADENOIDAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ALLERGIC GRANULOMATOUS ANGIITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 6 | 0
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHOSTENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 9 | 6
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 | 5
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 7
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 5 | 2
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 3
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY AMYLOIDOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 24 | 38
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PULMONARY INFARCTION (Respiratory, thoracic and mediastinal disorders) | 0 | 3
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CAPILLARITIS (Skin and subcutaneous tissue disorders) | 1 | 0
CUTANEOUS VASCULITIS (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 1
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 1 | 0
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 2
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 0 | 1
PURPURA (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 2
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1
PREGNANCY OF PARTNER (Social circumstances) | 1 | 0
ANGIODYSPLASIA (Vascular disorders) | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 0 | 1
AORTIC RUPTURE (Vascular disorders) | 0 | 1
ARTERIAL THROMBOSIS (Vascular disorders) | 1 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 2
DEEP VEIN THROMBOSIS (Vascular disorders) | 20 | 33
EMBOLISM VENOUS (Vascular disorders) | 2 | 0
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 0 | 1
HAEMATOMA (Vascular disorders) | 1 | 4
HYPERTENSION (Vascular disorders) | 1 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 2 | 0
HYPOTENSION (Vascular disorders) | 0 | 1
INTRA-ABDOMINAL HAEMATOMA (Vascular disorders) | 0 | 1
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 | 0
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 0 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 2 | 1
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 1
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 | 1
TEMPORAL ARTERITIS (Vascular disorders) | 1 | 0
THROMBOPHLEBITIS (Vascular disorders) | 0 | 3
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 0 | 2
VENA CAVA THROMBOSIS (Vascular disorders) | 0 | 1
VENOUS STENOSIS (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS (Vascular disorders) | 6 | 0
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=2676) | Enoxaparin/Warfarin (N=2689)
CONSTIPATION (Gastrointestinal disorders) | 73 | 87
DIARRHOEA (Gastrointestinal disorders) | 100 | 106
NAUSEA (Gastrointestinal disorders) | 81 | 106
VOMITING (Gastrointestinal disorders) | 50 | 69
FATIGUE (General disorders) | 58 | 50
OEDEMA PERIPHERAL (General disorders) | 93 | 111
PYREXIA (General disorders) | 54 | 56
BRONCHITIS (Infections and infestations) | 51 | 56
NASOPHARYNGITIS (Infections and infestations) | 104 | 98
URINARY TRACT INFECTION (Infections and infestations) | 92 | 82
CONTUSION (Injury, poisoning and procedural complications) | 48 | 97
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 30 | 105
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 33 | 78
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 38 | 56
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 28 | 55
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 74 | 84
BACK PAIN (Musculoskeletal and connective tissue disorders) | 80 | 87
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 119 | 130
DIZZINESS (Nervous system disorders) | 66 | 69
HEADACHE (Nervous system disorders) | 169 | 167
HAEMATURIA (Renal and urinary disorders) | 41 | 91
COUGH (Respiratory, thoracic and mediastinal disorders) | 61 | 58
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 64 | 73
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 77 | 144
HAEMATOMA (Vascular disorders) | 34 | 72
HYPERTENSION (Vascular disorders) | 70 | 68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.